CLINICAL TRIAL: NCT02100462
Title: Evaluation of Platelet Effects of Chlorthalidone and Hydrochlorothiazide
Brief Title: Chlorthalidone and HCTZ Impacts on Platelet Activation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Creighton University (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 13-16785
Record Dates: First submitted 2014-03-27; First posted 2014-04-01 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension
Keywords: Hypertension; Platelet activation; Platelet aggregation; Chlorthalidone
MeSH Terms: conditions — Hypertension | interventions — Chlorthalidone; Hydrochlorothiazide; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Chlorthalidone 12.5 mg (Experimental): Chlorthalidone 12.5 mg by mouth once daily for 2 weeks
  Interventions: Drug: Chlorthalidone 12.5 mg
- Hydrochlorothiazide 25 mg (Experimental): Hydrochlorothiazide 25 mg by mouth once daily for 2 weeks
  Interventions: Drug: Hydrochlorothiazide 25 mg
- Aspirin 81 mg (Active Comparator): Aspirin 81 mg by mouth once daily for 2 weeks
  Interventions: Drug: Aspirin 81 mg

INTERVENTIONS:
Drug: Chlorthalidone 12.5 mg
  Arms: Chlorthalidone 12.5 mg
Drug: Hydrochlorothiazide 25 mg
  Arms: Hydrochlorothiazide 25 mg
Drug: Aspirin 81 mg
  Arms: Aspirin 81 mg

SUMMARY:
This will be a randomized, double-blinded, three-period crossover study of platelet activation and aggregation in 30 non-smoking healthy volunteers comparing chlorthalidone (CTD), hydrochlorothiazide (HCTZ), and aspirin (ASA; active control). The study hypothesis is that CTD has different effects on platelet activation and aggregation than HCTZ.

ELIGIBILITY:
Inclusion Criteria:

* Men or women age 19 or older
* Not currently taking any routinely scheduled prescription or over the counter medications or herbal supplements
* No use of aspirin, clopidogrel, prasugrel, ticagrelor, cilostazol, dipyridamole, NSAID medications, or herbal supplements within the previous 7 days and able to refrain from use during the study period
* Systolic blood pressure > 110 mmHg and diastolic blood pressure > 60 mmHg
* Non-smoker

Exclusion Criteria:

* Previous adverse reaction or allergy to HCTZ, CTD, or ASA
* Severe sulfonamide hypersensitivity (anaphylaxis or Stevens-Johnson syndrome)
* Diagnosis of any chronic disease or condition
* History of gout or hyperuricemia
* History of pancreatitis
* History of systemic lupus erythematosus (SLE)
* History of hypokalemia requiring treatment
* Pregnant or planning to become pregnant during the study period
* Breastfeeding
* History of hypotension
* History of gastrointestinal bleeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Change in mean fluorescence intensity of PAC-1 | 2 weeks
  The primary endpoint for this study will be the change in mean fluorescence intensity (MFI) of the platelet activation marker PAC-1 due to HCTZ, CTD, and aspirin.

SECONDARY OUTCOMES:
Change in CD62P expression | 2 weeks
  Change in platelet expression of CD62P (p-selectin) in response to CTD, HCTZ, and ASA.
Change in platelet aggregation | 2 weeks
  Change in platelet aggregation measured by flow cytometry in response to CTD, HCTZ, and ASA

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Bashir, MD, Principal Investigator — Creighton University
Locations (1):
- Creighton University, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Bashir K, Burns T, Pirruccello SJ, Aurit SJ, Hilleman DE. Comparative antiplatelet effects of chlorthalidone and hydrochlorothiazide. J Clin Hypertens (Greenwich). 2022 Oct;24(10):1310-1315. doi: 10.1111/jch.14564. Epub 2022 Sep 6. PMID 36067089